CLINICAL TRIAL: NCT00198575
Title: A Multicenter, Prospective Cohort Study to Determine the Prevalence and Profile of Heparin-Induced Thrombocytopenia in Patients Undergoing Cardiovascular Surgery or Percutaneous Coronary Intervention
Brief Title: A Study on the Prevalence of Heparin-Induced Thrombocytopenia in Cardiovascular Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Other Study IDs: 15C-1-3
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2006-02

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: heparin-induced thrombocytopenia; cardiovascular surgery; percutaneous coronary intervention

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Several clinical studies in Western countries have revealed that the prevalence of HIT is 0.5 to 5%, varying depending on the clinical setting. Thirty to 50% of HIT patients suffer from thromboembolic events, and the mortality of HIT is 10 to 20%. In contrast, many physicians in Japan report no experience in treating HIT, although approximately 200,000 patients per year receive heparin. This raises the possibility that the prevalence of HIT might be much lower in Japan than in Western countries. In fact, neither the drug for HIT treatment nor the laboratory test for HIT diagnosis has been approved by the Pharmaceutical Affairs Law in Japan. We have therefore conducted a multi-center, prospective cohort study to determine the prevalence and profile of HIT in patients undergoing cardiovascular surgery or percutaneous coronary intervention. Approximately 1,500 patients will be enrolled in this study.

DETAILED DESCRIPTION:
Heparin is an important anticoagulation treatment, especially for cardiovascular patients. Recently, heparin-induced thrombocytopenia type II (HIT) has been shown to be an immune-mediated, life-threatening side effect of heparin therapy. Antibodies against heparin-platelet factor 4 (HIT antibodies), induced by heparin administration, are the major cause of HIT. HIT antibodies can stimulate platelets and endothelial cells, resulting in an excess production of thrombin, inducing thrombocytopenia and thromboembolic events. HIT typically occurs 5 to 14 days after the initial administration of heparin (typical-onset). HIT antibodies are transient but can be detected for about 100 days after the cessation of heparin treatment. Thus, some patients develop HIT either days after discontinuing heparin (delayed-onset) or soon after the re-administration of heparin (rapid-onset). HIT is clinically diagnosed by a drop in platelet count to less than 100,000/μL or a 50% decrease in platelets after the initiation of heparin therapy with no apparent explanation other than HIT. A positive laboratory test for HIT antibodies supports the clinical diagnosis.

Several clinical studies in Western countries have revealed that the prevalence of HIT is 0.5 to 5%, varying depending on the clinical setting. Thirty to 50% of HIT patients suffer from thromboembolic events, and the mortality of HIT is 10 to 20%. In contrast, many physicians in Japan report no experience in treating HIT, although approximately 200,000 patients per year receive heparin. This raises the possibility that the prevalence of HIT might be much lower in Japan than in Western countries. In fact, neither the drug for HIT treatment nor the laboratory test for HIT diagnosis has been approved by the Pharmaceutical Affairs Law in Japan. We have therefore conducted a multi-center, prospective cohort study to determine the prevalence and profile of HIT in patients undergoing cardiovascular surgery or percutaneous coronary intervention. Approximately 1,500 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females who meet the criteria listed below:

  1. Patients who are >=20 years of age
  2. Patients scheduled to undergo cardiovascular surgery or patients with acute coronary syndrome scheduled to undergo percutaneous coronary intervention
  3. Patients willing and able to give informed consent

Exclusion Criteria:

1. Patients who have a documented history of heparin-induced thrombocytopenia
2. Chronic thrombocytopenia (<100,000/μL)
3. Hematopoietic malignancy
4. Patients who receive an anticancer drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-11; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Miyata, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (13):
- Japan (13):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Hospital Organization Hakodate National Hospital, Hakodate, Hokkaido
  - Kurume University Hospital, Kurume, Hukuoka
  - Kobe City General Hospital, Kobe, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - National Cardiovascular Center, Suita, Osaka
  - Sakakibara Memorial Hospital, Fuchū, Tokyo
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni, Yamaguchi